CLINICAL TRIAL: NCT06198023
Title: Targeting Social Function to Improve Outcomes in Anxiety and Eating Disorders
Brief Title: Targeting Social Function in Anxiety and Eating Disorders
Acronym: SF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Carrie McAdams, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-1157
Record Dates: First submitted 2023-12-07; First posted 2024-01-10 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Atypical Anorexia Nervosa; Purging (Eating Disorders); Other Specified Feeding or Eating Disorder; Social Anxiety Disorder; Generalized Anxiety Disorder (GAD)
Keywords: social function; social cognition; social processing; psychoeducation; group therapy; group intervention; art therapy; social anxiety
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Phobia, Social; Generalized Anxiety Disorder; Social Adjustment | interventions — Drug Interactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Educational (Experimental)
  Interventions: Behavioral: Educational
- Interactive (Experimental)
  Interventions: Behavioral: Interactive

INTERVENTIONS:
Behavioral: Educational — The educational intervention is an 8-session series of informational presentations about brain function and altered social processing related to eating disorders. Participants will receive a reflective prompt to complete as homework and will have an opportunity to discuss their responses during the following session.
  Arms: Educational
Behavioral: Interactive — The interactive intervention is an 8-session series of experiential art therapy tasks followed by education about social processing. Participants will complete the tasks as a group or in small teams. Afterward, they will be encouraged to discuss their thoughts and feelings related to their experience. The educational component will include a homework assignment that participants will have the opportunity to discuss at the following session.
  Arms: Interactive

SUMMARY:
Social processing and cognition are often altered in patients with eating disorders. The goal of this clinical trial is to assess two different social therapeutic interventions -- one educational, one interactive -- for their effectiveness in improving clinical outcomes in patients with eating disorders. Patients in both interventions will receive education about social function in eating disorders, but those in the interactive treatment group will complete an additional collaborative art task.

Participants will:

* attend a baseline study visit to complete clinical interviews, cognitive testing, and behavioral tasks
* complete a pre-intervention assessment with questionnaires
* attend eight sessions of their assigned treatment group over the course of 12 weeks
* complete three virtual follow-up assessments 4, 8, and 12 months from their baseline
* attend a final study visit to repeat some clinical interviews, cognitive testing, and behavioral tasks

Researchers will compare changes in eating disorder, mood, and anxiety symptoms as well as test results from baseline and final study visits for each group to see if

* patients can be treated effectively with education alone or if an interactive group component produces additional benefits
* cognitive and behavioral task performance are associated with recovery or illness state.

DETAILED DESCRIPTION:
Eating disorders are devastating psychiatric disorders that afflict approximately 2% of young women and men. While the specific determining factors in illness progression and recovery remain poorly understood, social environment is known to be closely associated with eating disorders. Onset occurs most commonly in adolescence and young adulthood, times of complex changes in social roles, and social stressors are common both when eating disorders begin and recur. These clinical observations suggest that the brain mechanisms that process social stimuli may differ for people with eating disorders and therefore serve as powerful therapeutic targets. A previous interventional pilot targeting social function in eating disorders through psychoeducation and experiential tasks produced clinical improvements in the patients enrolled. This project will extend those results to evaluate whether the benefits experienced by participants are related to the therapeutic group interaction or can be achieved with education alone. Enrollment will be expanded to include males and individuals with OSFED (Other Specified Feeding and Eating Disorder) diagnoses. Additionally, to improve understanding of eating disorder course of illness, clinical symptoms, psychosocial behaviors, and neuropsychological function will be assessed at baseline and one year later.

Study Overview:

1. Group assignment will be determined based on time of study entry. Enrollment will alternate between interventions once researchers have recruited enough patients to fill a cohort (8-12 people).
2. Participants will attend an in-person baseline study visit to complete clinical interviews, neuropsychological testing, and computerized behavioral tasks.
3. Baseline self-report questionnaires will be completed virtually by participants prior to the first intervention session.
4. Both programs will consist of 8 sessions conducted across 12 weeks. This spacing allows for seasonal flexibility and accommodation of group member needs in order to maximize participation.
5. For participants in the educational arm, all intervention sessions will be completed remotely. Participants in the interactive will attend in-person sessions consisting of an hour-long art activity followed by the same hour-long psychoeducation session received by participants in the educational arm. Participants in both groups will be given homework assignments to complete after each session and invited to discuss their responses in the following session.
6. Participants will complete self-report questionnaires at time points T=4, 8, and 12, measured from the time of their baseline assessment. The T4 follow-up will include an evaluation form to collect participant feedback for the purpose of improving future interventions. Participants will also be asked to provide updates regarding their treatment, weight, medication(s), and similar information in a brief phone call with researchers.
7. After completing their T12 follow-up assessment, participants will attend a final in-person study visit to repeat some of the clinical, neuropsychological, and behavioral measures collected at baseline.

Participants who are unable or unwilling to complete their assigned intervention course will still be invited to complete follow-up assessments and a final study visit. This data will be valuable to the study's aim of better understanding the evolution of eating disorders over time.

ELIGIBILITY:
Inclusion Criteria:

* In the past 12 months, has met DSM-5 criteria met for an eating disorder (Anorexia Nervosa, Atypical Anorexia Nervosa, Bulimia Nervosa, Avoidant-Restrictive Food Intake Disorder, or Other Specified Feeding or Eating Disorder) and/or an anxiety disorder (Generalized Anxiety Disorder, Social Anxiety Disorder)
* Between the ages of 18-30

Exclusion Criteria:

* Current inpatient or residential treatment
* Medical instability or safety/suicide risk as determined by the PI

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in eating disorder symptoms | pre-intervention (T0) to four months from start of intervention (T4)
  The Eating Disorder Examination Questionnaire (EDE-Q) measures the severity of eating disorder symptoms. Possible scores on global eating disorder pathology range from 0 to 6, with higher scores indicating greater severity. Scores of 2 or less are considered typical of normative eating behavior/cognitions, while scores of 3-6 suggest the presence of clinically significant eating disorder symptoms.
Change in eating disorder symptoms | four months from start of intervention (T4) to eight months from start of intervention (T8)
  The Eating Disorder Examination Questionnaire (EDE-Q) measures the severity of eating disorder symptoms. Possible scores on global eating disorder pathology range from 0 to 6, with higher scores indicating greater severity. Scores of 2 or less are considered typical of normative eating behavior/cognitions, while scores of 3-6 suggest the presence of clinically significant eating disorder symptoms.
Change in eating disorder symptoms | eight months from start of intervention (T8) to twelve months from start of intervention (T12)
  The Eating Disorder Examination Questionnaire (EDE-Q) measures the severity of eating disorder symptoms. Possible scores on global eating disorder pathology range from 0 to 6, with higher scores indicating greater severity. Scores of 2 or less are considered typical of normative eating behavior/cognitions, while scores of 3-6 suggest the presence of clinically significant eating disorder symptoms.
Change in eating disorder symptoms | pre-intervention (T0) to twelve months from start of intervention (T12)
  The Eating Disorder Examination Questionnaire (EDE-Q) measures the severity of eating disorder symptoms. Possible scores on global eating disorder pathology range from 0 to 6, with higher scores indicating greater severity. Scores of 2 or less are considered typical of normative eating behavior/cognitions, while scores of 3-6 suggest the presence of clinically significant eating disorder symptoms.
Change in depression symptoms | pre-intervention (T0) to four months from start of intervention (T4)
  The Patient Health Questionnaire (PHQ-9) is a 9-item measure of depression symptoms. Each item is rated on a four-point scale (0 = not at all; 1 = several days; 2 = more than half the days; 3 = nearly every day). Possible scores range from 0-27, allowing depression to be categorized as minimal (1-4), mild (5-9), moderate (10-14), moderately severe (15-19), or severe (20-27).
Change in depression symptoms | four months from start of intervention (T4) to eight months from start of intervention (T8)
  The Patient Health Questionnaire (PHQ-9) is a 9-item measure of depression symptoms. Each item is rated on a four-point scale (0 = not at all; 1 = several days; 2 = more than half the days; 3 = nearly every day). Possible scores range from 0-27, allowing depression to be categorized as minimal (1-4), mild (5-9), moderate (10-14), moderately severe (15-19), or severe (20-27).
Change in depression symptoms | eight months from start of intervention (T8) to twelve months from start of intervention (T12)
  The Patient Health Questionnaire (PHQ-9) is a 9-item measure of depression symptoms. Each item is rated on a four-point scale (0 = not at all; 1 = several days; 2 = more than half the days; 3 = nearly every day). Possible scores range from 0-27, allowing depression to be categorized as minimal (1-4), mild (5-9), moderate (10-14), moderately severe (15-19), or severe (20-27).
Change in depression symptoms | pre-intervention (T0) to twelve months from start of intervention (T12)
  The Patient Health Questionnaire (PHQ-9) is a 9-item measure of depression symptoms. Each item is rated on a four-point scale (0 = not at all; 1 = several days; 2 = more than half the days; 3 = nearly every day). Possible scores range from 0-27, allowing depression to be categorized as minimal (1-4), mild (5-9), moderate (10-14), moderately severe (15-19), or severe (20-27).
Change in anxiety symptoms | pre-intervention (T0) to four months from start of intervention (T4)
  The General Anxiety Disorder Scale (GAD-7) is a 7-item measure of anxiety symptoms. Each item is rated on a four-point scale (0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day). Possible scores range from 0-21, allowing anxiety to be classified as minimal (0-4), mild (5-9), moderate (10-14), or severe (15-21).
Change in anxiety symptoms | four months from start of intervention (T4) to eight months from start of intervention (T8)
  The General Anxiety Disorder Scale (GAD-7) is a 7-item measure of anxiety symptoms. Each item is rated on a four-point scale (0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day). Possible scores range from 0-21, allowing anxiety to be classified as minimal (0-4), mild (5-9), moderate (10-14), or severe (15-21).
Change in anxiety symptoms | eight months from start of intervention (T8) to twelve months from start of intervention (T12)
  The General Anxiety Disorder Scale (GAD-7) is a 7-item measure of anxiety symptoms. Each item is rated on a four-point scale (0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day). Possible scores range from 0-21, allowing anxiety to be classified as minimal (0-4), mild (5-9), moderate (10-14), or severe (15-21).
Change in anxiety symptoms | pre-intervention (T0) to twelve months from start of intervention (T12)
  The General Anxiety Disorder Scale (GAD-7) is a 7-item measure of anxiety symptoms. Each item is rated on a four-point scale (0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day). Possible scores range from 0-21, allowing anxiety to be classified as minimal (0-4), mild (5-9), moderate (10-14), or severe (15-21).
Change in overall levels of psychopathology | pre-intervention (T0) and at the last post-intervention follow-up (T12)
  The DSM-5 Cross-Cutting Symptom Measure (DSM-XC) is a 23-item measure of overall levels of psychopathology across 13 psychiatric domains. Each item on the measure is rated on a 5-point scale (0=none or not at all; 1=slight or rare, less than a day or two; 2=mild or several days; 3=moderate or more than half the days; and 4=severe or nearly every day). The score on each item within a domain should be reviewed. Because additional inquiry is based on the highest score on any item within a domain, the clinician is asked to indicate that score in the "Highest Domain Score" column
Change in eating disorder diagnosis | baseline and final study visits (approximately 1 year apart)
  The Eating Disorder Diagnostic Assessment for DSM-5 (EDA-5) is a semi-structured clinical interview meant to assist in the assessment of a feeding or eating disorder according to DSM-5 criteria.

SECONDARY OUTCOMES:
Change in verbal learning and memory | baseline and final study visits (approximately 1 year apart)
  California Verbal Learning Test (CVLT-3) is an individually administered assessment that measures both recall and recognition of two lists of words over a number of immediate and delayed memory trials. The CVLT 3 Core Report contains demographics, a core score summary, a scaled score profile, a standard score summary, a process score summary, and demographically adjusted core and standard scores, if selected. Item responses for all recall trials can also be selected for inclusion on the report.
Change in visuospatial learning and memory | baseline and final study visits (approximately 1 year apart)
  Ruff-Light Trail Learning Test (RULIT) is a measure of visuospatial learning and memory. The respondent is given a stimulus card containing a complex configuration of circles interconnected by lines and asked to use an index finger to trace a line connecting the circles from the START to the END. The task is repeated until participants trace the correct path in two consecutive trials. Immediate Memory is assessed by the number of steps correctly completed in Trial 2. Learning is assessed by the number of trials to master the task and the cumulative number of errors across Trials 2 through 10 (or until the task is mastered), and Long-term Recall is evaluated by having the respondent retrace the trail after a 60-minute delay.
Change in sense of social connectedness | pre-intervention (T0) to four months from start of intervention (T4)
  The Social Connectedness Scale (SCS) is a self-report questionnaire that measures the extent to which individuals feel connected to others in their social environment. It consists of 20 items that assess four different dimensions of social connectedness that include belongingness, closeness, support, and satisfaction. Individuals rate each item on a 6-point Likert scale, from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate a greater sense of social connectedness.
Change in sense of social connectedness | four months from start of intervention (T4) to eight months from start of intervention (T8)
  The Social Connectedness Scale (SCS) is a self-report questionnaire that measures the extent to which individuals feel connected to others in their social environment. It consists of 20 items that assess four different dimensions of social connectedness that include belongingness, closeness, support, and satisfaction. Individuals rate each item on a 6-point Likert scale, from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate a greater sense of social connectedness.
Change in sense of social connectedness | eight months from start of intervention (T8) to twelve months from start of intervention (T12)
  The Social Connectedness Scale (SCS) is a self-report questionnaire that measures the extent to which individuals feel connected to others in their social environment. It consists of 20 items that assess four different dimensions of social connectedness that include belongingness, closeness, support, and satisfaction. Individuals rate each item on a 6-point Likert scale, from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate a greater sense of social connectedness.
Change in sense of social connectedness | pre-intervention (T0) to twelve months from start of intervention (T12)
  The Social Connectedness Scale (SCS) is a self-report questionnaire that measures the extent to which individuals feel connected to others in their social environment. It consists of 20 items that assess four different dimensions of social connectedness that include belongingness, closeness, support, and satisfaction. Individuals rate each item on a 6-point Likert scale, from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate a greater sense of social connectedness.
Change in perceived social support | pre-intervention (T0) to four months from start of intervention (T4)
  The Multidimensional Scale of Perceived Social Support is a 12-item measure of perceived adequacy of social support from three sources -- family, friends, & significant other -- using a 5-point Likert scale (0 = strongly disagree, 5 = strongly agree).
Change in perceived social support | four months from start of intervention (T4) to eight months from start of intervention (T8)
  The Multidimensional Scale of Perceived Social Support is a 12-item measure of perceived adequacy of social support from three sources -- family, friends, & significant other -- using a 5-point Likert scale (0 = strongly disagree, 5 = strongly agree).
Change in perceived social support | eight months from start of intervention (T8) to twelve months from start of intervention (T12)
  The Multidimensional Scale of Perceived Social Support is a 12-item measure of perceived adequacy of social support from three sources -- family, friends, & significant other -- using a 5-point Likert scale (0 = strongly disagree, 5 = strongly agree).
Change in perceived social support | pre-intervention (T0) to twelve months from start of intervention (T12)
  The Multidimensional Scale of Perceived Social Support is a 12-item measure of perceived adequacy of social support from three sources -- family, friends, & significant other -- using a 5-point Likert scale (0 = strongly disagree, 5 = strongly agree).
Change in trait self-esteem | pre-intervention (T0) to four months from start of intervention (T4)
  Rosenberg trait self-esteem Scale (TSE) is a 10-item measure of global self-worth. Each item is rated on a four-point Likert scale from (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree) and five items are reverse scored. Higher scores indicate higher self-esteem.
Change in trait self-esteem | four months from start of intervention (T4) to eight months from start of intervention (T8)
  Rosenberg trait self-esteem Scale (TSE) is a 10-item measure of global self-worth. Each item is rated on a four-point Likert scale from (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree) and five items are reverse scored. Higher scores indicate higher self-esteem.
Change in trait self-esteem | eight months from start of intervention (T8) to twelve months from start of intervention (T12)
  Rosenberg trait self-esteem Scale (TSE) is a 10-item measure of global self-worth. Each item is rated on a four-point Likert scale from (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree) and five items are reverse scored. Higher scores indicate higher self-esteem.
Change in trait self-esteem | pre-intervention (T0) to twelve months from start of intervention (T12)
  Rosenberg trait self-esteem Scale (TSE) is a 10-item measure of global self-worth. Each item is rated on a four-point Likert scale from (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree) and five items are reverse scored. Higher scores indicate higher self-esteem.
Change in social learning rates | baseline to final study visit (approximately 1 year apart)
  Cyberball is is an online ball-tossing game that participants believe they are playing with three others. In the version we are using, one player (good) preferentially includes the participant, one (neutral) is equitable, and another player (bad) stops throwing the ball to the participant. Changes in the percentage of throws to each type of player indicate responsivity to social learning. The percentage of throws to the good player will increase while the percentage of throws to the bad player will decrease as participants become more attuned to valence of social interactions.
Change in social reward learning | baseline to final study visit (approximately 1 year apart)
  The Trust Game is a tend-round economic game in which two players take turns acting as "investor" and "trustee." The investor is given $20 and sends a portion to the trustee. The trustee receives three times the invested amount and returns some amount to the investor. This task provides total amounts earned; larger amounts indicate more attunement to the partner's behavior. We hypothesize that this will increase after the intervention due to improved sensitivity to others.
Change in social learning biases | baseline to final study visit (approximately 1 year apart)
  The Evaluation Learning Task presents participants with 6 computer personas across two conditions (self-referential or other-referential). Participants are given word pairs (e.g. 'witty' vs. 'dull') and are asked to guess which word the computer persona would use to describe them (SR) or 'George' (OR). Using the feedback on their selections (correct or incorrect), they must decide whether the computer persona liked or disliked them and to what degree (%). Participant response times and proportion of correct responses in each condition (like, neutral, or dislike) are used to evaluate learning rates and biases in each condition.
Change in attribution biases | baseline to final study visit (approximately 1 year apart)
  The Causal Attribution Task measures latent tendency to attribute positive and negative everyday events to internal (vs external) and global (vs specific) causes.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie J McAdams, MD PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Multispecialty Psychiatry Clinic, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryan A, Arthur S, Lieu L, Kallianpur R, Mahmood F, Noebel N, Sherman-Chung M, McAdams CJ. Learning to connect: feasibility, acceptability and experiences in the social domain intervention for eating disorders. J Eat Disord. 2025 Nov 23;13(1):294. doi: 10.1186/s40337-025-01470-0. PMID 41276826